CLINICAL TRIAL: NCT03044106
Title: The Effects of Cranial Laser Reflex Technique on Hamstring Flexibility, Strength, and Pain Pressure Threshold: a Pilot Study
Brief Title: Cranial Laser Reflex Technique for Hamstring Function
Acronym: CLRTHam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0898
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2017-10

CONDITIONS: Hamstring Injury; Muscle Tone Increased; Muscle Pain; Muscle Weakness
Keywords: hamstrings; flexibility; strength; pain pressure threshold; lllt; photobiomodulation; cranial reflex; cranial laser reflex technique; CLRT
MeSH Terms: conditions — Muscle Hypertonia; Myalgia; Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Subjects who meet the inclusion criteria and give consent were randomized to one of the following for the first treatment period: 1) active CLRT; or 2) sham laser. At the first intervention visit, the research assistant entered the subject's assigned identification into an online computer program (selected by study biostatistician) to determine assignment to one of the two periods. The study biostatistician used computer-generated random numbers to generate the allocation sequence using random blocks of random sizes. A one-week washout period minimized carryover effects.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects and assessors were blinded to treatment allocation. The subject was face down, eyes closed, and wearing protective eyewear that blocks the specific wavelength of the laser light during the intervention.
  After each treatment session, the participants completed a de-blinding questionnaire administrated by the assessor providing a dichotomous 'yes' or 'no' answer as to whether active treatment was received. This response was followed by a second question regarding how certain they were that active treatment was received on a 0-10 numeric rating scale (NRS), where 0 represents absolutely uncertain and 10 represents absolutely certain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CLRT, Then Sham (Active Comparator): Subjects performed the KEA, HHD, PPT functional tests on their right hamstring before and after the CLRT intervention.
  Interventions: Device: CLRT
- Sham, Then CLRT (Sham Comparator): The Sham procedure was identical to CLRT except the laser device was placed in placebo mode: all device indicator lights and sounds will be functional but no laser light will be emitted from probe aperture.
  Interventions: Device: CLRT

INTERVENTIONS:
Device: CLRT — CLRT is a novel method of laser stimulation on specific cranial reflex points that modulate muscle tone.
  Other Names: Cranial Laser Reflex Technique

SUMMARY:
Purpose: To conduct a pilot study of the effect of Cranial Laser Reflex Technique (CLRT) compared with sham laser on hamstring muscle flexibility, strength, and pain pressure threshold.

Participants: Active, young adults ages 18 to 35.

Procedures: A two-visit, assessor and participant-blinded crossover study with 1-week washout. Subjects will complete three functional hamstring tests before and after CLRT and sham laser treatment. Subjects will also complete questionnaires to assess their expectations and perceptions of the interventions.

DETAILED DESCRIPTION:
First Visit: Subjects who met the inclusion criteria and gave consent completed a brief questionnaire on their activity level, history of hamstring injuries, and perceived hamstring tightness and were randomized to one of the following for the first treatment period: 1) active CLRT; or 2) sham laser.

After randomization, subjects were asked to complete the three functional hamstring tests: 90-90 Knee Extension Angle (KEA) to assess flexibility, handheld dynamometry (HHD) for strength, and pain pressure threshold (PPT).

Assessments. KEA: The 90-90 Knee Extension Angle test is a functional assessment designed to assess lower extremity flexibility and is considered the gold standard for hamstring length. The participant began in the supine position on a treatment table. The tested extremity (the right leg in each subject) was placed in a 90° hip and 90° knee position with the contralateral lower extremity placed flat on the table. A digital inclinometer was consistently placed at the level of the medial malleoli and the superior pole of the patella. The examiner maintained 90° of hip flexion. Pelvic position was monitored by palpation of the anterior superior iliac spine and lumbar spinous processes to maintain a neutral pelvic position. The examiner passively extended the knee to the point of a ''strong, but tolerable stretch," as reported by the subject. The examiner read the angle of the inclinometer and recorded the mean value of three attempts. A greater angle indicates greater degree of flexibility.

Hand held Dynamometry (HHD) is currently considered a reliable and valid measurement of peak muscle contraction. The subject began prone on the table with right leg bent to 90°. The tester placed the dynamometer (microFET2; Hoggan Health Industries, Salt Lake City, UT) at the heel of the participant and applied force to the heel, gradually increasing in 3 to 5 seconds. Participants was instructed to resist the applied force and maximally contract the hamstring muscle against the HHD device. The test ended once they are no longer able to resist the force and the leg begins to move (break point). The investigator recorded the mean value of three attempts.

Pain Pressure Threshold (PPT) is a reliable, accurate and valid method for measuring muscle pain sensitivity and response to treatment. The digital algometer (FDX, Wagner Instruments, Greenwich, CT) is a hand-held muscle tester with a range of 0-100 lbf that consists of a padded disc with a diameter of 0.5" attached to a microprocessor-control unit that measures peak force (pounds or kilograms). The unit has a digital readout for peak-applied pressure and provides a built-in calibration routine that verifies a valid calibration. In order to determine PPT, the researcher applied the tip of the algometer to a tender spot in the participant's hamstrings and increased the amount of pressure until the participant verbally informed the researcher when the sensation of pressure became pain. At this point the algometer was removed and the peak force recorded. The mean of three repeated measures was reported.

Intervention: Cranial Laser Reflex Technique (CLRT) is a novel complementary and alternative (CAM) medicine intervention for musculoskeletal conditions that incorporates principles of laser acupuncture with chiropractic cranial reflexology. Subjects wore protective eyewear. The hamstring reflexes are two lines on the posterior portion of the top of the head, approximately 2 cm long and 2 cm apart, running parallel to the sagittal suture. The posterior end of the reflexes can be located by finding the vertex, or CZ point in the standardized 10-20 EEG system, and moving laterally approximately 1 cm.

The aperture of the laser probe was placed at the posterior end of the reflex (b), turned on and moved anteriorly to point (a) at a speed of approximately 2 cm/s. The laser was turned off and quickly returned to the starting point, turned on and moved again. This was repeated for a total of 30 times. The probe skimmed the surface of the scalp, moving aside as much hair as possible.

Device: The treatment device used in this study is a Class IIIB 810nm 200 milliwatts (mW) near-infrared diode laser (THOR Photomedicine Ltd, Great Britain) that is currently marketed in the US. The laser probe is FDA-cleared and classified as a non-significant risk device. The spot size is 0.0364 cm^2, and the treatment time is 30 seconds. Current best-practice recommendations for laser acupuncture recommend a dosage between 1-4 J/cm^2 per point. Since the CRP is a line of 2 cm, for the purposes of calculating dosage, it was treated as a series of 10 connected points each with a diameter of 2mm. With the scanning rate of 2cm/s, each "point" on the line received 1/10 of each pass, totaling 3s (out of 30s total) exposure time per point. The dose per point for this intervention is calculated to be approximately 1.65 J/cm^2.

There was a one-week washout and the subject will return for the second treatment period.

Primary Outcome: Hamstring flexibility (90-90 Knee Extension Angle, KEA) A clinically significant effect size is an increase of 5 degrees. The investigator recorded the mean value of three attempts. Hypothesis: CLRT will increase hamstring flexibility.

Secondary Outcomes:

1. Hamstring Strength as assessed by Handheld Dynamometry. HHD . The investigator recorded the mean value of three attempts. Hypothesis: CLRT will have a neutral to positive effect on hamstring strength.
2. Pain Pressure Threshold. The mean of three repeated measures was reported. An increase in PPT signifies an increase in pain tolerance. Hypothesis: CLRT will increase pain tolerance.
3. Age, gender, activity level, perceived hamstring tightness, perceived hamstring flexibility and perceived hamstring strength were assessed at baseline and subsequent follow up visit. Results were stratified by these variables to assess interaction with treatment.

Sample Size and Power: Based on previously published results, a mean increase of 5º on the KEA (e.g., from 135º to 140º) is considered to be clinically meaningful, assuming a common standard deviation of 15º. It is also assumed that correlation between repeated measurements from the same individual will be at least 0.75 (likely a conservative assumption). Under these assumptions, enrolling 38 participants would provide at least 80% power using a two-sided test at the 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-35 years of age
2. All genders
3. Willing to complete two study visits over 2-3 weeks
4. Able to read and communicate in English

Exclusion Criteria:

1. Current lower back condition with pain, numbness or tingling that radiates down the legs
2. Active treatment for a major medical illness, such as heart disease, uncontrolled diabetes or hypertension, malignancy, autoimmune, or immune deficiency disorder
3. History of vasculitis, intracranial mass, clotting disorder (including medication-induced, e.g., warfarin)
4. Current skin malignancy on scalp
5. Cognitive dysfunction preventing informed consent
6. Pending or currently receiving benefits from personal injury litigation, including worker's compensation
7. Chronic long-term disability related to lumbosacral injury/symptoms
8. Epilepsy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Wise, D.C., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC- Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — https://clrtforhamstrings.web.unc.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- CLRT, Then SHAM: Subject will perform KEA (knee extension angle), HHD (handheld dynamometry), PPT (pain pressure threshold) functional tests. Investigator will record the mean of 3 attempts for each test. Subject will don protective eyewear. CLRT (Cranial Laser Reflex Technique) will be performed: the aperture of the laser probe will be placed at one end of the reflex (a), turned on and moved to the end of the reflex (b) at a speed of approximately 2 cm/s. The laser will be turned off and quickly returned to point (a), turned on and moved to point (b) again. This will be repeated for a total of 30 times. After CLRT is completed, the KEA, PPT and HHD tests will be repeated and the mean of 3 attempts for each will be recorded.
- SHAM, Then CLRT: The identical procedures will be followed as in the other arm. The only difference is the the laser device will be in sham mode: all lights and sounds are operational with no laser emission from the aperture.
Period: Visit 1
Arm/Group | CLRT, Then SHAM | SHAM, Then CLRT
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | CLRT, Then SHAM | SHAM, Then CLRT
Started | 22 | 22
Completed | 22 | 20
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Visit 2
Arm/Group | CLRT, Then SHAM | SHAM, Then CLRT
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: This is the total of all participants that began the trial and completed at least one visit.
Arm/Group | All Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.02 (3.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 38
  More than one race | 2
  Unknown or Not Reported | 0
Injury, either leg, last 6 months [Count of Participants; unit: Participants] | 4
surgery to either leg, ever [Number; unit: participants] | 5
Prior hamstring strain history [Count of Participants; unit: Participants] | 8
Subjective hamstring tightness [Count of Participants; unit: Participants]
  Very tight | 5
  Somewhat tight | 20
  A little tight | 11
  Not at all tight | 4
  Unknown | 4

OUTCOME MEASURES:

1. Primary Outcome: 90-90 Knee Extension Angle Test
Description: Knee Extension Angle (KEA) test is a functional test designed to assess lower extremity flexibility and is considered the gold standard test for assessing hamstring length. Results will be recorded as degrees of knee flexion angle. A clinically significant effect size is an increase of 5 degrees.
Time Frame: At baseline and immediately after intervention
Population: Analysis was conducted on intention to treat.
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- CLRT: Subject will don protective eyewear. The hamstring reflexes are two lines on the posterior portion of the top of the head. The treatment device to be used in this study is a Class 3B, 810 nanometer (nm), 200 milliwatt (mW) near-infrared diode laser (THOR Photomedicine Ltd, Great Britain) that is currently marketed in the US.The aperture of the laser probe will be placed at the posterior end of the reflex, turned on and moved to the anterior end of the reflex at a speed of approximately 2 cm/s. The laser will be turned off and quickly returned to point (a), turned on and moved to point (b) again. This will be repeated for a total of 30 times.
- SHAM: The Sham procedure will be identical to CLRT except the laser device will be in placebo mode: all device indicator lights and sounds will be functional but no laser light will be emitted from probe aperture.
Arm/Group | CLRT | SHAM
Number analyzed (Participants) | 42 | 44
degrees
  KEA at baseline/pre-intervention | 167.3 (8.4) | 166.4 (8.8)
  KEA immediately post-intervention | 168.5 (9.3) | 168.8 (7.5)

2. Secondary Outcome: Handheld Dynamometry
Description: Handheld Dynamometry (HHD) is measures peak muscle contraction. The measurements will be recorded as kilograms (kg) and higher scores indicate higher muscle strength. The subject will be prone on the table with right leg bent to 90° and will maximally contract the hamstring muscle for 4-5 seconds against the HHD device. The investigator will record the mean value of three attempts. Higher scores indicate greater strength.
Time Frame: At baseline and immediately after intervention
Population: Intention to treat.
Measure: Mean (Standard Deviation); unit: Kilograms
Groups:
- CLRT: Subject will don protective eyewear. The hamstring reflexes are two lines on the posterior portion of the top of the head. The aperture of the laser probe will be placed at the posterior end of the reflex (a), turned on and moved to the anterior end of the reflex (b) at a speed of approximately 2 cm/s. The laser will be turned off and quickly returned to point (a), turned on and moved to point (b) again. This will be repeated for a total of 30 times.
  The spot size is 0.0364 cm², and the treatment time is 30 seconds. Since the CRP is a line of 2 cm, for the purposes of calculating dosage, we will treat it as a series of 10 connected points each with a diameter of 2mm. With the scanning rate of 2 cm/s, each "point" on the line will receive 1/10 of each pass, totaling 3s (out of 30s total) exposure time per point. The dose per "point" for this intervention is calculated to be approximately 1.65 J/cm².
Arm/Group | CLRT | Sham
Number analyzed (Participants) | 42 | 44
Kilograms
  HHD at baseline/pre-intervention | 17.2 (4.7) | 17.4 (4.6)
  HHD immediately post-intervention | 16.9 (4.5) | 17.0 (4.7)

3. Secondary Outcome: Pain Pressure Threshold
Description: PPT is a reliable, accurate and valid method for measuring muscle pain sensitivity and response to treatment. In order to determine PPT, the researcher will apply the tip of the algometer to a tender spot in the participant's hamstrings and increase the amount of pressure until the participant verbally informs the researcher when the sensation of pressure became pain. At this point the algometer is removed and the peak force recorded. The mean of three repeated measures will be reported. An increase in PPT signifies an increase in pain tolerance and a decrease in pain sensitivity.
Time Frame: At baseline and immediately after intervention
Population: Intention to treat.
Measure: Mean (Standard Deviation); unit: kgf
Groups:
- CLRT: Subject will don protective eyewear. The hamstring reflexes are two lines on the posterior portion of the top of the head. The aperture of the laser probe will be placed at the posterior end of the reflex (a), turned on and moved to the anterior end of the reflex (b) at a speed of approximately 2 cm/s. The laser will be turned off and quickly returned to point (a), turned on and moved to point (b) again. This will be repeated for a total of 30 times.
  The spot size is 0.0364 cm², and the treatment time is 30 seconds. Since the CRP is a line of 2 cm, for the purposes of calculating dosage, we will treat it as a series of 10 connected points each with a diameter of 2mm. With the scanning rate of 2cm/s, each "point" on the line will receive 1/10 of each pass, totaling 3s (out of 30 s total) exposure time per point. The dose per "point" for this intervention is calculated to be approximately 1.65 J/cm².
Arm/Group | CLRT | Sham
Number analyzed (Participants) | 42 | 44
kgf
  PPT at baseline/pre-intervention | 10.6 (3.6) | 11.0 (3.9)
  PPT immediately post-intervention | 11.3 (4.6) | 11.5 (4.5)

4. Secondary Outcome: Mean Difference Pre/Post KEA, Stratified by History of Prior Hamstring Strain
Description: Mean difference between active CLRT and Sham in hamstring flexibility (KEA) stratified by a history of prior hamstring injury. 8 participants reported prior injuries, 36 reported having no prior hamstring strain.
Time Frame: At baseline and immediately after intervention
Population: Mean difference in pre/post KEA after receiving active CLRT and Sham in hamstring flexibility (KEA), stratified by a history of prior hamstring injury.
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Active CLRT, History of Hamstring Strain: Participants receiving active treatment who reported a prior history of hamstring strain (n=8). This group approximates a clinical population.
- Sham CLRT With History of Hamstring Strain: Participants receiving sham treatment who reported a prior history of hamstring strain (n=8)
- Active CLRT With no Prior Hamstring Strain: Participants receiving active treatment who reported no prior history of hamstring strain (n=36)
- Sham CLRT With no History of Hamstring Strain: Participants receiving sham CLRT with no history of hamstring strain
Arm/Group | Active CLRT, History of Hamstring Strain | Sham CLRT With History of Hamstring Strain | Active CLRT With no Prior Hamstring Strain | Sham CLRT With no History of Hamstring Strain
Number analyzed (Participants) | 8 | 8 | 36 | 36
degrees
  PRE KEA | 167.825 (7.925141) | 168.4875 (8.898384) | 167.1778 (8.58657) | 165.9235 (8.778143)
  POST KEA | 171.65 (6.762501) | 169.4875 (8.092225) | 167.8417 (9.658316) | 168.6118 (7.420887)
Statistical Analysis 1: Comparison: Active CLRT, History of Hamstring Strain; This is the difference between pre and post KEA in those receiving the active treatment with a history of hamstring strain; Test type: Superiority; p = 0.0068, t-test, 2 sided; Mean Difference (Final Values) = 3.825, 95% CI 2-sided [1.058809 to 6.591192], Standard Deviation 3.308759
Statistical Analysis 2: Comparison: Sham CLRT With History of Hamstring Strain; This is the difference in pre /post KEA means after receiving the sham treatment in those with a history of hamstring strains; Test type: Superiority; p = 0.2185, t-test, 2 sided; Median Difference (Final Values) = 1.0, 95% CI 2-sided [-1.869044 to 3.869044], Standard Deviation 3.431784
Statistical Analysis 3: Comparison: Active CLRT With no Prior Hamstring Strain; This is the difference in pre/post KEA means in those receiving the active treatment with no history of hamstring strain; Test type: Superiority; p = 0.1281, t-test, 2 sided; Mean Difference (Final Values) = .6638904, 95% CI 2-sided [-.5037233 to 1.831504], Standard Deviation 3.450892
Statistical Analysis 4: Comparison: Sham CLRT With no History of Hamstring Strain; This is the difference in pre/post KEA means in those receiving the sham treatment who have no history of hamstring strain; Test type: Superiority; p = 0.00, t-test, 2 sided; Mean Difference (Final Values) = 2.688237, 95% CI 2-sided [1.557137 to 3.819337], Standard Deviation 3.241751
Statistical Analysis 5: Comparison: Active CLRT, History of Hamstring Strain vs Sham CLRT With History of Hamstring Strain; This is the mean difference in effect between active and sham in those with a history of hamstring strain; Test type: Superiority; p = 0.090, Mixed Models Analysis; Mean Difference (Final Values) = 2.825, 95% CI 2-sided [-0.4543 to 6.0581]
Statistical Analysis 6: Comparison: Active CLRT With no Prior Hamstring Strain vs Sham CLRT With no History of Hamstring Strain; This is the mean difference of effect between active and sham in those without a history of hamstring strain; Test type: Superiority; p = 0.018, Mixed Models Analysis; Mean Difference (Final Values) = -2.024, 95% CI 2-sided [-3.4474 to -0.3406]

ADVERSE EVENTS:
Time Frame: Data was collected on two visits separated by at least 1 week washout period. On the second visit, participants were asked about any adverse events. A survey on adverse events was sent 2 weeks after second visit asking for any information on adverse everts as well.
Groups:
- CLRT: Subject will don protective eyewear. The hamstring reflexes are two lines on the posterior portion of the top of the head. The aperture of the laser probe will be placed at posterior end of the reflex (a), turned on and moved to the anterior end of the reflex (b) at a speed of approximately 2 cm/s. The laser will be turned off and quickly returned to point (a), turned on and moved to point (b) again. This will be repeated for a total of 30 times.
- SHAM: The laser is inactive, all other descriptions are the same as active.
Arm/Group | CLRT | SHAM
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 1/44 | 2/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLRT (N=44) | SHAM (N=44)
Mild soreness in Hamstring (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Mild Headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The high baseline flexibility of the population may have a ceiling effect on the intervention. Further examination of the effects of CLRT in a clinical population is warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT03044106/Prot_SAP_000.pdf